CLINICAL TRIAL: NCT01498510
Title: Web-based CBT for Opioid-treated, Chronic Pain Patients With Aberrant Behavior
Brief Title: Web-based Cognitive-behavior Therapy (CBT) for Opioid-treated, Chronic Pain Patients With Aberrant Behavior
Acronym: WebCBTPain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Development and Research Institutes, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WebCBTPain618; R01DA026887 (NIH)
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Chronic Pain
Keywords: chronic pain; cognitive behavior therapy; web-based intervention
MeSH Terms: conditions — Chronic Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment-as-usual (TAU) (No Intervention): The standard medical treatment provided to chronic pain patients at the study site pain specialty practice
- TAU plus web-based intervention (Experimental): An interactive, web-based intervention, based on principles of cognitive behavior therapy (CBT), that teaches chronic pain patients with aberrant behavior self-management skills to reduce pain severity and medication misuse and improve functioning
  Interventions: Behavioral: Web-based CBT for chronic pain

INTERVENTIONS:
Behavioral: Web-based CBT for chronic pain — An interactive, web-based intervention, based on principles of cognitive behavior therapy (CBT), that is designed to train chronic pain patients in self-management skills to reduce pain and aberrant behavior and improve functioning
  Other Names: cognitive behavior therapy (CBT); web-based intervention
  Arms: TAU plus web-based intervention

SUMMARY:
The purpose of this study is to develop and evaluate an innovative, web-based self-management intervention for opioid-treated chronic pain patients who display aberrant drug-related behavior.

DETAILED DESCRIPTION:
Within the past decade, there has been increasing recognition of the limitations and risks of opioid therapy for chronic pain, spurred by the U.S.' widespread epidemic of opioid misuse. Within the clinical context, concerns about long-term opioid therapy persist due to limited evidence of efficacy and the occurrence of medication misuse/abuse (termed aberrant drug-related behavior). Psychosocial approaches, particularly self-management strategies such as cognitive-behavior therapy (CBT), have been found to be efficacious for the treatment of chronic pain. However, most chronic pain patients are not exposed to comprehensive psychosocial interventions, due to factors including pain specialty physicians' lack of familiarity with and time to provide behavioral treatments and insufficient payer coverage for these therapies. To address these public health concerns, this study developed, implemented and evaluated an innovative, web-based CBT intervention for the treatment of chronic pain tailored to the specific needs of patients who are prescribed opioids and present with aberrant behavior. The development of this interactive, web-based intervention was informed by iterative feedback from pain experts and chronic pain patients. In a randomized, controlled trial, chronic pain patients receiving opioid therapy at a pain specialty practice were assigned to receive 12 weeks of either treatment-as-usual (TAU; n=55) or treatment-as-usual plus the web-based intervention (Web-CBT; n=55). The trial evaluated the relative effectiveness of these treatments on the primary outcomes of pain severity, pain interference and aberrant opioid-taking behavior, and the secondary outcomes of pain catastrophizing and pain-related Emergency Department visits. Additional analyses explored the impact of the intervention on several supplementary outcomes, such as various categories of activities, psychiatric distress and positive affect, and examined hypothesized mediators of treatment outcome, including quality of life, social support and expectations about the future.

ELIGIBILITY:
Inclusion Criteria:

* moderate-to-severe pain for at least 3 months (score of 5 or greater on Brief Pain Inventory)
* patient at pain treatment program study site
* prescribed opioid analgesics
* aberrant drug-related behavior within the past 30 days (endorsing 4 or more items on the Current Opioid Misuse Measure)

Exclusion Criteria:

* primary headache or cancer pain
* scheduled for major surgery within the next 6 months
* described by physician as likely to die within the next year
* plans to move out of the area within the next 3 months
* insufficient ability to provide informed consent or insufficient English to participate in consent process, assessments or computer intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-02; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
pain severity, as measured by the Multidimensional Pain Inventory (MPI) | 6 months
pain interference, as measured by the Multidimensional Pain Inventory (MPI) | 6 months
aberrant drug-related behavior, assessed via the Current Opioid Misuse Measure (COMM) | 6 months

SECONDARY OUTCOMES:
pain catastrophizing, measured by the Pain Catastrophizing Scale (PCS) | 6 months
Emergency Department visits for pain | 6 months

OTHER OUTCOMES:
General Activities, Social Activities, Activities Away from Home, Household Chores | 6 months
  activity sub-scales of the Multidimensional Pain Inventory (MPI)
psychiatric distress, assessed via the SCL-10R | 6 months
positive affect, assessed by the Positive Affect Negative Affect Scale (PANAS) | 6 months
quality of life, as measured by the World Health Organization Quality of Life-BREF | 6 months
social support, assessed by the MOS Social Support Scale | 6 months
expectations about the future, assessed by the Future Scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Rosenblum, Ph.D., Principal Investigator — National Development and Research Institutes, Inc.; Lisa A. Marsch, Ph.D., Principal Investigator — Dartmouth College
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided